CLINICAL TRIAL: NCT01262625
Title: ACRIN-4701 RESCUE: Randomized Evaluation of Patients With Stable Angina Comparing Utilization of Diagnostic Examinations
Brief Title: Randomized Evaluation of Patients With Stable Angina Comparing Diagnostic Examinations
Acronym: RESCUE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding timeline completed
Sponsor: American College of Radiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ACRIN 4701 RESCUE; 1R01HS019403 (AHRQ)
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Results first posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Chest Pain; Stable Angina Pectoris, CCS Class I to III; Angina Equivalent; Coronary Artery Disease
Keywords: stable angina; recurrent chest pain; chest pain; angina equivalent; diagnosis; coronary artery disease
MeSH Terms: conditions — Chest Pain; Angina, Stable; Coronary Artery Disease; Disease | interventions — Exercise Test; Tomography, Emission-Computed, Single-Photon; Myocardial Perfusion Imaging

STUDY DESIGN:
Intervention Model Description: This randomized, controlled, diagnostic, multicenter trial will follow participants at 6-month intervals for up to 24 months to determine the incidence of MACE, defined as myocardial infarction (MI) or cardiac-related death, and cross-over to revascularization.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A: CCTA Diagnostic (Experimental): Participants randomized to diagnostic evaluation using coronary computed tomographic angiography (CCTA) to determine therapeutic course of action.
  Interventions: Device: CCTA
- Group B: SPECT MPI/ICA Diagnostic (Active Comparator): Standard-of-care diagnostic assessment using single photon emission computed tomography myocardial perfusion imaging (SPECT MPI), possibly followed by diagnostic invasive coronary angiography (ICA) dependent on SPECT MPI results.
  Interventions: Device: SPECT MPI/ICA

INTERVENTIONS:
Device: CCTA — Complete diagnostic CCTA per protocol specifications.
  Other Names: coronary CT; cardiac CT; coronary computed tomographic angiography
  Arms: Group A: CCTA Diagnostic
Device: SPECT MPI/ICA — Perform SPECT MPI per institutional standard practice; diagnostic ICA will be performed only as indicated per protocol.
  Other Names: nuclear medicine cardiac stress test; stress test; nuclear medicine stress test; cardiac stress test; exercise cardiac stress test; pharmacologic cardiac stress test; single photon emission computed tomography (SPECT) myocardial perfusion imaging (MPI)
  Arms: Group B: SPECT MPI/ICA Diagnostic

SUMMARY:
This randomized, controlled, diagnostic, multicenter trial will compare two diagnostic imaging pathways--coronary computed tomography angiography (CCTA) and single photon emission tomography (SPECT) myocardial perfusion imaging (MPI)--to determine the incidence of major adverse coronary events (MACE), defined as myocardial infarction (MI) or cardiac-related death, and cross-over to revascularization. CCTA may be used to direct patients with symptoms of stable angina or angina equivalent to optimal medical therapy (OMT). The use of CCTA as a diagnostic tool for angina symptoms will be associated with no increase in MACE or revascularization, decreased cost, reduced risks (e.g., less radiation exposure), additional insights into alternate explanations of chest pain, and increased cost-effectiveness in comparison with use of SPECT MPI/invasive coronary angiography (ICA).

DETAILED DESCRIPTION:
The Randomized Evaluation of Patients with Stable Angina Comparing Utilization of Diagnostic Examinations (RESCUE) is a multi-center randomized, controlled trial responding to the need for comparative analysis of these imaging technologies and the role of OMT in clinical care. A total of 4300 patients will be randomized to CCTA or SPECT MPI/ICA for diagnostic assessment of angina at up to 80 institutions internationally. This study builds on the results of the COURAGE trial by comparing CCTA and SPECT MPI/ICA integrated into a care paradigm featuring initial treatment with OMT for patients diagnosed using computer-aided diagnosis (CAD) without significant disease in the left main coronary artery. Participants will be followed for a composite endpoint of MACE and cross-over to revascularization over a follow-up period up to two years (two to six time points depending on diagnostic results and time of enrollment into the trial). The primary endpoint of the study is a combined endpoint of occurrence of MACE and revascularization. We will calculate differences in the combined MACE/revascularization endpoint between the CCTA and SPECT MPI/ICA arms. Participant outcomes will be assessed by age, gender, comorbidity, and angina classification class at presentation. Several comparative-effectiveness analyses will be performed. We hypothesize that the CCTA arm will be associated with no increase in MACE or revascularization, decreased cost, reduced risks (e.g., less radiation exposure), additional insights into or alternate explanations of chest pain, and increased cost-effectiveness in comparison with SPECT MPI/ICA. Findings are expected to result in validation of an evolving new standard of care for patients with stable angina that takes advantage of CCTA and OMT to more cost-effectively drive appropriate care while reducing the need for invasive diagnosis and increased radiation exposure with SPECT MPI/ICA.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide a written informed consent;
* 40 years or older;
* Presentation with symptoms of stable angina (CCS Class I to III) or angina equivalent with or without known CAD;
* Planned non-invasive imaging for CAD diagnosis;
* Able to tolerate CCTA or SPECT MPI per randomization as required by protocol, to be performed at an ACRIN-qualified facility with a RESCUE-qualified scanner.

Exclusion Criteria:

* Prior revascularization;
* Not suitable to undergo CT with an iodinated contrast agent:

  * Known allergy-like reaction to contrast media as defined by the American College of Radiology (ACR) (see www.acr.org/SecondaryMainMenuCategories/quality_safety/contrast_manual.aspx for reaction definition) or moderate to severe allergic reactions to more than one allergen;
  * Renal failure, as determined by glomerular filtration rate (GFR) < 30 mL/min/1.73 m2 based on a serum creatinine level obtained within 28 days prior to registration;
* Renal insufficiency at the time of enrollment, as determined by GFR 30 to 60 mL/min/1.73 m2 based on a serum creatinine level obtained within 28 days prior to registration, unless permitted by the institution's policy and/or ACR guidance for risk reduction strategies (see www.acr.org/SecondaryMainMenuCategories/quality_safety/contrast_manual.aspx for guidance on contrast selection and pre-treatment strategies);
* Atrial fibrillation or significant arrhythmia judged to potentially limit quality of CCTA;
* Acute ischemia;
* Acute myocardial infarction;
* Severe myocardial ischemia: known markedly positive exercise treadmill stress test (ST) [significant ST segment depressions or hypotensive response during stage I of the Bruce protocol];
* Unable to suspend respiration for 15 seconds or to follow instructions to do so;
* Unstable angina and symptoms refractory to maximal oral and intravenous medical therapy (persistent CCS Class IV);
* History of known left ventricular ejection fraction < 45%;
* Pulmonary edema or heart failure unresponsive to standard medical therapy;
* Pacemaker;
* Valvular heart disease likely to require surgery in the next 18 months;
* Congenital heart disease or cardiomyopathy likely to affect prognosis during follow up;
* Significant systemic hypertension (blood pressure > 200/100 mm Hg) unresponsive to medical therapy;
* Severe noncardiovascular comorbidity limiting survival (e.g., cancer or other life threatening illness for which the patient is expected to live less than 12 months);
* Prior imaging evaluation for this episode of symptoms (e.g., SPECT MPI or CCTA within the previous 72 hours);
* BMI > 40 kg/m2;
* Pregnancy or intent to become pregnant (if a female is of childbearing potential-defined as a premenopausal female capable of becoming pregnant-a pregnancy test should be done prior to enrollment).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2011-05-20 (Actual); Primary Completion 2014-11-26 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Stillman, MD, PhD, Principal Investigator — Division of Cardiothoracic Imaging, Emory University; Pamela K Woodard, MD, Study Chair — Mallinckrodt Institute of Radiology, Washington University of Medicine
Locations (3):
- United States (3):
  - Atlantic VA Medical Center, Decatur, Georgia
  - Henry Ford Hospital, Detroit, Michigan
  - Salem VA Medical Center, Salem, Virginia

REFERENCES:
- [Background] Boden WE, O'Rourke RA, Teo KK, Hartigan PM, Maron DJ, Kostuk WJ, Knudtson M, Dada M, Casperson P, Harris CL, Chaitman BR, Shaw L, Gosselin G, Nawaz S, Title LM, Gau G, Blaustein AS, Booth DC, Bates ER, Spertus JA, Berman DS, Mancini GB, Weintraub WS; COURAGE Trial Research Group. Optimal medical therapy with or without PCI for stable coronary disease. N Engl J Med. 2007 Apr 12;356(15):1503-16. doi: 10.1056/NEJMoa070829. Epub 2007 Mar 26. PMID 17387127
- [Background] Shaw LJ, Berman DS, Maron DJ, Mancini GB, Hayes SW, Hartigan PM, Weintraub WS, O'Rourke RA, Dada M, Spertus JA, Chaitman BR, Friedman J, Slomka P, Heller GV, Germano G, Gosselin G, Berger P, Kostuk WJ, Schwartz RG, Knudtson M, Veledar E, Bates ER, McCallister B, Teo KK, Boden WE; COURAGE Investigators. Optimal medical therapy with or without percutaneous coronary intervention to reduce ischemic burden: results from the Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation (COURAGE) trial nuclear substudy. Circulation. 2008 Mar 11;117(10):1283-91. doi: 10.1161/CIRCULATIONAHA.107.743963. Epub 2008 Feb 11. PMID 18268144
- [Derived] Stillman AE, Gatsonis C, Lima JAC, Liu T, Snyder BS, Cormack J, Malholtra V, Schnall MD, Udelson JE, Hoffmann U, Woodard PK; RESCUE investigators *. Coronary Computed Tomography Angiography Compared With Single Photon Emission Computed Tomography Myocardial Perfusion Imaging as a Guide to Optimal Medical Therapy in Patients Presenting With Stable Angina: The RESCUE Trial. J Am Heart Assoc. 2020 Dec 15;9(24):e017993. doi: 10.1161/JAHA.120.017993. Epub 2020 Dec 5. PMID 33283579

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to enrollment in May 2011 and was closed to enrollment in June 2013 due to resource limitations.
  The study was designed to enroll and randomize 4300 participants to the 2 study arms, but given the difficulties of recruiting enough patients to fulfill the stringent entry criteria, as well as time constraints for funding (American Recovery and Reinvestment Act award, 3-year cap), only one quarter of the planned sample size could be recruited .
Period: Overall Study
Arm/Group | Group A: CCTA Diagnostic | Group B: SPECT MPI/ICA Diagnostic
Started | 518 | 532
Scan Available | 475 | 465
Uninterpretable Scan | 6 | 4
Completed | 516 | 531
Not Completed | 2 | 1
Not completed — Administrative Error | 1 | 1
Not completed — Site Closed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: CCTA Diagnostic: Participants randomized to diagnostic evaluation using CCTA to determine therapeutic course of action.
  CCTA: Complete diagnostic CCTA per protocol specifications.
- Group B: SPECT MPI/ICA Diagnostic: Standard-of-care diagnostic assessment using SPECT MPI, possibly followed by diagnostic ICA dependent on SPECT MPI results.
  SPECT MPI/ICA: Perform SPECT MPI per institutional standard practice; diagnostic ICA will be performed only as indicated per protocol.
- Total: Total of all reporting groups
Arm/Group | Group A: CCTA Diagnostic | Group B: SPECT MPI/ICA Diagnostic | Total
Number analyzed (Participants) | 516 | 531 | 1047
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9) | 58 (9) | 58 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233 | 244 | 477
  Male | 283 | 287 | 570
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 58 | 104
  Not Hispanic or Latino | 467 | 468 | 935
  Unknown or Not Reported | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 7 | 15
  Asian | 11 | 14 | 25
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 73 | 77 | 150
  White | 400 | 415 | 815
  More than one race | 10 | 5 | 15
  Unknown or Not Reported | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Time-dependent Rates of the Composite Primary Endpoint Major Adverse Cardiovascular Event (MACE: Comprising Cardiac-related Death or Acute Myocardial Infarction (AMI), and Revascularization)
Description: To compare outcomes of participants with symptoms of stable angina or angina equivalent evaluated with an anatomic imaging strategy using CCTA as initial method of computer-aided diagnosis (CAD) (Group A) to a combined functional and anatomic imaging strategy of SPECT MPI/ICA (Group B) as a guide to Optimal Medical Therapy (OMT) alone.
  The analysis was conducted from an intent-to-treat perspective
Time Frame: up to 24 Months (depends on time of trial enrollment and funding duration)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: CCTA Diagnostic | Group B: SPECT MPI/ICA Diagnostic
Number analyzed (Participants) | 516 | 531
Participants
  No Event | 487 | 504
  Event Occurred | 29 | 27
Statistical Analysis 1: Comparison: Group A: CCTA Diagnostic vs Group B: SPECT MPI/ICA Diagnostic; Test type: Non-Inferiority or Equivalence — the pre-defined non-inferiority margin of 1.25; p = 0.19, Regression, Cox; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.61 to 1.75]

2. Secondary Outcome: Prediction of Response (MACE/Revascularization) at 1 Year Using: Modified Duke Score or CCTA + AHA 16 Predictor/CCTA+AHA 16+Clinical Data Predictor or SPECT% Reversible Defect Size Reported as Receiver Operating Characteristic (ROC) Area Under Curve (AUC)
Description: AUC is a unitless measure of performance ranging form 0.5 (guessing) to 1.0 (perfect predictor) that can be thought of a the proportion of correct classifications in a 2-alternative-forced-choice experiment - and for binary outcomes, it is equivalent to the C-statistic.
  It will be used to evaluate and compare the ability of available prognostic indices and SPECT-MPI % reversible defect size to predict revascularization or MACE using CCTA information:
  A CCTA Modified Duke index A CCTA index including the 16 individual American Heart Association (AHA) segments A CCTA including the 16 individual AHA segments and clinical data and compare them to the SPECT % reversible defect size results
Time Frame: 1 year
Population: For the secondary analyses, patients with <1-year follow-up (defined as <335 days) were excluded from analysis, as were ineligible patients and patients without the respective randomized scan or with an uninterpretable scan The analysis will compare the the proposed SPECT % reversible defect size vs the a modified Duke Score and the standard CCTA +AHA 16 to predict MACE events.
Measure: Number (95% Confidence Interval); unit: unitless
Groups:
- Group A: CCTA Modified Duke Score: The modified Duke prognostic CAD index was calculated as outlined by Min & colleagues (Min et al 2007) for Group A CCTA Participants
- Group A: CCTA + AHA 16 Predictor: A new predictive model based upon the raw CCTA stenosis data using the AHA 16-segments: graded as normal (0%), very mild (1-29%), mild (30-49%), moderate (50-69%), or severe (≥70%) stenosis for Group A CCTA Participants. Because of the relatively few MACE events, these were grouped to <30%, 30-49%, and ≥50% for subsequent analysis.
- Group A: CCTA + AHA 16 + Clinical Data Predictor: A new predictive model based upon the raw CCTA stenosis data using the AHA 16-segments: graded as normal (0%), very mild (1-29%), mild (30-49%), moderate (50-69%), or severe (≥70%) stenosis for Group A CCTA Participants. Because of the relatively few MACE events, these were grouped to <30%, 30-49%, and ≥50% for subsequent analysis.
  Hypertension was included in the model as the only clinical risk factor selected by multivariate modeling.
- Group B: SPECT % Reversible Defect Size: Standard-of-care (SOC) diagnostic assessment using SPECT MPI (Group B)
  % Reversible defect size calculated as per institutional SOC.
Arm/Group | Group A: CCTA Modified Duke Score | Group A: CCTA + AHA 16 Predictor | Group A: CCTA + AHA 16 + Clinical Data Predictor | Group B: SPECT % Reversible Defect Size
Number analyzed (Participants) | 401 | 401 | 401 | 378
unitless | 0.87 [0.81 to 0.94] | 0.92 [0.87 to 0.96] | 0.93 [0.89 to 0.97] | 0.73 [0.59 to 0.88]
Statistical Analysis 1: Comparison: Group A: CCTA Modified Duke Score vs Group B: SPECT % Reversible Defect Size; Test type: Superiority; p = 0.08, DeLong; (DeLong et al 1988)
Statistical Analysis 2: Comparison: Group A: CCTA + AHA 16 Predictor vs Group B: SPECT % Reversible Defect Size; Test type: Superiority; p = 0.02, DeLong; (DeLong et al 1988)

3. Secondary Outcome: Short Form-36 Survey (SF-36v2) and Seattle Angina Questionnaire (SAQ) Score
Description: SF36+SAQ at baseline and to a subset of participants, stratified by diagnostic examination, at 12 months after enrollment to monitor angina symptoms and their impact on Quality of life.
  The Short Form-36 (SF36) is a 36 item overall health status/Quality of Life collected in 8 domains. Scales are standardized with scores ranging from 0-100. Higher scores= better health status.
  The Seattle Angina Questionnaire (SAQ) is a self-administered, 19-item, cardiac disease-related quality-of-life measure collected in 5 domains. scales are standardized with scores ranging from 0-100. Higher scores= better health status.
  Positive cardiac findings on diagnostic testing are defined as:
  1. 50% stenosis on CCTA or un-evaluable left main, or proximal and mid segments of all other epicardial arteries (right coronary artery, left anterior descending artery, or left circumflex artery); and
  2. 10% reversible defect on SPECT MPI or evidence of Transient Ischemic Dilation (TID) accompanied by ECG
Time Frame: baseline and 12 months
Population: Only cases with and an available screen result and both baseline and 1-year surveys completed are included in this analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Group A: CCTA Diagnostic - Negative; Group A: CCTA Diagnostic - Positive: Participants randomized to diagnostic evaluation using CCTA to determine therapeutic course of action.
  A positive case is defined as 50% stenosis on CCTA or un-evaluable left main, or proximal and mid segments of all other epicardial arteries (right coronary artery, left anterior descending artery, or left circumflex artery);
- Group B: SPECT MPI/ICA Diagnostic - Negative; Group B: SPECT MPI/ICA Diagnostic - Positive: Standard-of-care diagnostic assessment using SPECT MPI, possibly followed by diagnostic ICA dependent on SPECT MPI results.
  SPECT MPI/ICA: Perform SPECT MPI per institutional standard practice; diagnostic ICA will be performed only as indicated per protocol.
  a positive case is defined as having a 10% reversible defect on SPECT MPI or evidence of TID accompanied by ECG changes of ischemia.
Arm/Group | Group A: CCTA Diagnostic - Negative | Group B: SPECT MPI/ICA Diagnostic - Negative | Group A: CCTA Diagnostic - Positive | Group B: SPECT MPI/ICA Diagnostic - Positive
Number analyzed (Participants) | 132 | 155 | 42 | 10
score on a scale
  SF-36: Phys comp: Baseline | 45.41 (9.27) | 46.07 (9.69) | 46.10 (8.51) | 47.2 (9.19)
  SF-36: Phys Func: Baseline | 46.41 (10.48) | 47.16 (9.98) | 46.4 (9361) | 46.3 (12.37)
  SF-36: Role-physical: Baseline | 46.07 (10.22) | 46.76 (10.26) | 45.77 (8.79) | 48.04 (10.07)
  SF36: Bodily pain: Baseline | 45.83 (9.11) | 45.87 (8.72) | 46.31 (7.94) | 45.55 (9.65)
  SF36: General health: Baseline | 47.10 (9.01) | 46.43 (9.51) | 46.17 (8.13) | 50.31 (5.08)
  SF36: Mental comp: Baseline | 49.42 (11.15) | 48.52 (10.64) | 47.09 (9.55) | 49.46 (6.91)
  SF36: Vitality: Baseline | 48.11 (10.23) | 46.75 (10.9) | 47.9 (9.86) | 46.75 (10.90)
  SF36: Social functioning: Baseline | 46.60 (10.63) | 47.25 (10.42) | 46.86 (9.40) | 49.76 (5.17)
  SF36: Role emotional: Baseline | 47.9 (12.07) | 48.08 (11.12) | 44.96 (10.16) | 48.51 (9.77)
  SF36: Mental health: Baseline | 49.98 (10.16) | 48.51 (9.77) | 47.83 (9.36) | 50.01 (7.39)
  SAQ: Physical limitation: Baseline | 67.50 (15.83) | 67.12 (17.20) | 65.20 (16.67) | 67.41 (17.36)
  SAQ: Angina stability: Baseline | 44.34 (31.42) | 48.87 (32.71) | 40.98 (30.32) | 38.00 (27.41)
  SAQ: Angina frequency: Baseline | 77.38 (15.24) | 79.79 (15.40) | 74.25 (16.15) | 75.00 (15.81)
  SAQ: Treatment satisfaction: Baseline | 84.64 (15.57) | 85.87 (15.95) | 85.85 (15.41) | 82.94 (11.91)
  SAQ: Disease perception: Baseline | 58.74 (20.18) | 59.33 (19.81) | 54.38 (19.06) | 62.50 (19.74)
  SF36: Physical component: 1-Year | 47.44 (10.66) | 46.39 (10.4) | 47.27 (8.66) | 52.51 (5.04)
  SF36: Physical functioning: 1-Year | 46.96 (10.77) | 47.35 (10.46) | 46.56 (9.31) | 51.77 (5.97)
  SF36: Role-physical: 1-Year | 48.14 (11.28) | 46.00 (11.07) | 48.38 (9.20) | 53.42 (4.65)
  SF36: Bodily pain: 1-Year | 47.96 (10.15) | 46.62 (10.16) | 45.91 (10.13) | 53.03 (7.14)
  SF36: General health: 1-Year | 49.10 (10.74) | 46.40 (10.86) | 46.84 (9.84) | 53.55 (7.64)
  SF36: Mental comp: 1-Year | 50.11 (10.82) | 48.11 (10.96) | 46.69 (11.50) | 53.51 (6.93)
  SF36: Vitality: 1-Year | 50.09 (40.51) | 47.78 (11.49) | 48.72 (11.15) | 53.96 (6.45)
  SF36: Social functioning: 1-Year | 48.72 (11.15) | 53.96 (6.45) | 48.54 (10.77) | 46.72 (11.21)
  SF36: Role emotional: 1-Year | 48.43 (11.07) | 46.89 (11.59) | 46.25 (9.84) | 52.38 (7.87)
  SF36: Mental health: 1-Year | 50.17 (10.24) | 48.26 (10.38) | 46.45 (11.58) | 54.23 (6.40)
  SAQ: Physical limitation: 1-Year | 71.98 (16.65) | 68.80 (17.83) | 66.61 (17.39) | 76.30 (10.77)
  SAQ: Angina stability: 1-Year | 80.31 (28.17) | 82.52 (27.26) | 71.71 (30.98) | 92.00 (19.32)
  SAQ: Angina frequency: 1-Year | 92.46 (11.36) | 92.59 (14.71) | 86.00 (16.46) | 97.00 (6.75)
  SAQ: Treatment satisfaction: 1-Year | 87.40 (17.89) | 86.85 (20.74) | 84.90 (18.42) | 97.65 (3.04)
  SAQ: Disease perception: 1-Year | 79.03 (20.16) | 77.58 (21.77) | 71.04 (23.64) | 91.67 (13.61)

4. Secondary Outcome: The Effectiveness of Each Arm Will be Measured in Terms of Life Years and Quality of Life Years (QALY).
Description: International medical records will be used to determine mortality which may not be feasible at all participating international sites.
  Utilities will be based on Quality of Well Being scores converted from the SF-36 assessments The analysis will be performed assuming a societal perspective and lifetime time horizon
Time Frame: Baseline and 1 year
Population: The study was terminated before data to compute life years was collected SF-36 scores have been reported previously
Arm/Group | Group A: CCTA Diagnostic | Group B: SPECT MPI/ICA Diagnostic
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 day after Imaging
Arm/Group | Group A: CCTA Diagnostic | Group B: SPECT MPI/ICA Diagnostic
All-Cause Mortality (participants affected / at risk) | 0/518 | 0/532
Serious Adverse Events (participants affected / at risk) | 0/518 | 0/532
Other Adverse Events (participants affected / at risk) | 0/518 | 0/532

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2011-05-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT01262625/Prot_SAP_ICF_000.pdf